CLINICAL TRIAL: NCT05819645
Title: Early Versus Delayed Oral Fluid Intake Initiation (Sipping) After Extubation, Influence on the Feeling of Thirst, Patient Comfort and the Occurrence of Complications.
Brief Title: Oral Fluid Intake After Extubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Durila Miroslav MUDr. Ph.D., prf., University Hospital, Motol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK-1381/22
Record Dates: First submitted 2023-01-06; First posted 2023-04-19 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early fluid intake (Experimental)
  Interventions: Behavioral: Fluid intake not as per standard guidlines
- Standard Delayed oral fluid (Other)
  Interventions: Behavioral: Fluid intake not as per standard guidlines

INTERVENTIONS:
Behavioral: Fluid intake not as per standard guidlines — The participant will be randomized into two arms. After the randomization one arm will get the per os fluid intake before the standard time frame.

SUMMARY:
According to the current guidelines the patient is not allowed to drink any fluid at least 2 hours after extubation to prevent complications. However there is no evidence in the literature to support this approach. Because anaesthetic drugs and their side effects changed significantly from their first usage, the investigators can assume that existing approach is obsolete and has no place anymore in the modern medicine. Keeping patient n.p.o (nothing per os) for 2 hours after extubation may lead to patient´s thirst or other discomfort. The aim of the study is to detect whether early oral fluid intake after extubation could lead to safe relief of thirst and to better patient´s comfort overall.

DETAILED DESCRIPTION:
Everything stated in the brief summary.

ELIGIBILITY:
Inclusion Criteria:

* patients with planned extubation assigned to the study
* able to swallow the fluid
* willing to participate the study

Exclusion Criteria:

* patients after upper digestive tract surgery
* patients after trachea surgery
* patients with possible neurological deficiency
* patients after VIII. cranial nerve surgery
* patients not able to swallow

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Assessment of presence or absence of thirst 120 minutes after extubation | During procedure (120 minutes after extubation)
  Between both groups the presence of anpleasent feeling of thirst will be assessed and compared

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Motol, Charles University in Prague, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sedlackova S, Nigrovicova V, Peckova M, Durila M. Immediate "sipping" vs. delayed oral fluid intake after extubation: A randomized controlled trial. J Crit Care. 2026 Feb;91:155212. doi: 10.1016/j.jcrc.2025.155212. Epub 2025 Aug 7. PMID 40780083